CLINICAL TRIAL: NCT03701880
Title: The Impact of Ivabradine Administration on Clinical Outcome and Biomarkers of Decompensated Heart Failure
Brief Title: Early Use of Ivabradine in Heart Failure
Acronym: Ivabradine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Sadat City University (Other)
Responsible Party: Principal Investigator, Nouran Ahmed Aly, Teaching Assistant of Clinical Pharmacy department, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ClinicalPH110
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Decompensated Heart Failure
Keywords: Decompensated Heart Failure; Ivabradine; ST2 Biomarker
MeSH Terms: interventions — Ivabradine; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine group (Experimental): an initial dose of 5 mg/12 hours of Ivabradine will be added to beta-blockers (bisoprolol 2.5 mg/day) and ivabradine will be increased until a dose of 7.5 mg/12 hours according to HR. The heart rate target will be at least <70 bpm and not lower than 60 bpm. If HR decreases below 60 bpm, ivabradine and/or beta-blockers doses will be decreased to the previous dose. After discharge, beta-blockers up-titration will be continued during follow-up visit.
  Interventions: Drug: Ivabradine; Drug: Bisoprolol
- Control group (Active Comparator): beta-blocker (bisoprolol 2.5 mg/day) and it will be doubled every 2 weeks during the admission according to the stability of HR, blood pressure and tolerability of patients. Ivabradine will be only added after reaching bisoprolol optimal dose (10mg) or maximum tolerated dose and the HR is still above 70 bpm. If HR decreases below 60 bpm, ivabradine dose will be decreased.
  Interventions: Drug: Ivabradine; Drug: Bisoprolol

INTERVENTIONS:
Drug: Ivabradine — Ivabradine is pacemaker current I(f) inhibitor thereby slowing heart rates without exhibiting negative inotropic effect on the myocardium or altering ventricular action potential
  Other Names: Procoralan
Drug: Bisoprolol — Bisoprolol is beta-blocker
  Other Names: concor

SUMMARY:
The aim of the work is to Evaluate the efficacy, quality of life and safety of early addition of ivabradine to B-blocker in reduced EF heart failure patients after acute decompensation compared to the standard treatment.

DETAILED DESCRIPTION:
this study is a Prospective randomized open label study will be conducted on Egyptian patient with heart failure with reduced ejection fraction(rEF HF). Each of the eligible patients will be randomized to one of these groups, early administration of Ivabradine and B-blocker group or control group which follows American Heart Association treatment guidelines of rEF HF.

The objectives include the following:

1. Physical examination (heart rate, blood pressure, dyspnea and orthopnea symptoms)
2. NYHA class
3. Pro-NT-BNP serum level, ST2 serum level
4. Echocardiography (left ventricular ejection fraction)
5. Score of Minnesota Living with Heart Failure Questionnaire these objectives will be measured baseline, 2 weeks and after 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Patient with acute heart failure either newly diagnosed or decompensated heart failure after stabilization
2. Patients > 18 years old
3. Left ventricular ejection fraction less than 40 % of presumed irreversible etiology
4. Clinically stable 24-48 hours after admission
5. Sinus rhythm with heart rate above 70 bpm
6. No previous treatment with ivabradine

Exclusion Criteria:

1. Patients less than 18 years.
2. Arterial fibrillation before inclusion.
3. Ventricular dysfunction due to acute event (Myocarditis, AMI). 4- cardiogenic shock

5. Patients are taking drug interact with ivabradine. 6- carrier or candidate for pacemaker, heart transportation, cardiac surgery or other cardiovascular procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-16 (Actual); Primary Completion 2019-12-23 (Estimated); Study Completion 2019-12-23 (Estimated)

PRIMARY OUTCOMES:
serum Pro-BNP level | 3 months
  Elevated NT-proBNP parallel HF disease severity and it is suggestive of worse clinical outcomes and mortality in HF

SECONDARY OUTCOMES:
ST2 serum level | 3 months
  Repeated ST2 measurements appeared to be a strong predictor of outcome especially in patients with acute HF. Also, ST2 levels in patients with acute HF are significantly higher than in patients with chronic HF and fall rapidly over days to weeks during HF treatment. This lack of reduction in ST2 level during acute HF treatment is predictive of mortality. So, persistently high levels of ST2 were associated with increased mortality risk
The effect on patient quality of life using Minnesota Living with Heart Failure Questionnaire | 3 months of follow-up.
  The questionnaire is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. the patient marks a 0 (zero) to 5 scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. it is simply scored by summation of all 21 responses.The simple sum of the responses that ranges from 0 to 105 is a measurement of heart failure severity as indicated by its adverse effect on the respondent's life during the past month
NYHA class assessment | 3 months
  This classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath
Heart rate | 3 months
  Measuring heart rate
Left ventricular ejection fraction assessment | 3 months
  Two-dimensional echocardiogram coupled with Doppler flow studies will be performed
Blood pressure | 3 months
  Measuring systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- El Demerdash Hospital, Cairo, Egypt